CLINICAL TRIAL: NCT04234581
Title: The Effect of Lysulin on Glycemic Control and Advanced Glycation in Inadequately Controlled Type 2 Diabetes Mellitus: a Double Blinded Placebo Controlled Study
Brief Title: The Effect of Lysulin on Glycemic Control and Advanced Glycation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Juraj Koska (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Juraj Koska, Senior Research Health Scientist, Carl T. Hayden VA Medical Center
Organization: Carl T. Hayden VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1185
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes
Keywords: lysine; vitamin C; zinc; hemoglobin A1c; advanced glycation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lysulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lysulin (Experimental): Participants will be randomly allocated in blocks for 3 months to LysulinTM (1,110 mg TID, i.e. 3.3 g/day) per os with breakfast, lunch and dinner.
  Interventions: Dietary Supplement: Lysulin
- Placebo (Placebo Comparator): Subjects will be instructed to take two tablets of placebo per os with breakfast, lunch and dinner.
  Interventions: Dietary Supplement: Lysulin

INTERVENTIONS:
Dietary Supplement: Lysulin — Participants will be randomly allocated for 3 months to LysulinTM (1,110 mg TID, i.e. 3.3 g/day) or matching placebo.

SUMMARY:
The primary objective is to determine whether 12 weeks of treatment with Lysulin, compared to placebo, causes a reduction from baseline in the plasma levels of glucose, hemoglobin A1c (HbA1c) and Advanced Glycation Endproducts (AGEs) in patients with inadequately controlled type 2 diabetes mellitus. Secondary objectives include determining whether 12 weeks of treatment with Lysulin increases beta-cell function as measured by plasma C-peptide levels.

DETAILED DESCRIPTION:
Objective(s): The primary objective is to determine whether 12 weeks of treatment with Lysulin, compared to placebo, causes a reduction from baseline in the plasma levels of glucose, hemoglobin A1c (HbA1c) and Advanced Glycation Endproducts (AGEs) in patients with inadequately controlled type 2 diabetes mellitus. Secondary objectives include determining whether 12 weeks of treatment with Lysulin increases beta-cell function as measured by plasma C-peptide levels.

Research Plan: A randomized, prospective, double-blind study with randomization to lysulin and placebo in a 1:1 fashion. The study will enroll 60 patients with inadequately controlled type 2 diabetes.

Methods: The study will be performed as outpatient study at Phoenix VA Clinical Research Center. The study will include 3-4 visits. At the initial visit, participants will complete informed consent proc HbA1c ≥ 7.5 % and < 10%ess and undergo screening examination. Inclusion criteria will be age 21-75 years, HbA1c ≥ 7.5 % and < 10%, and stable dose of insulin 6 weeks prior to enrollment. Qualified participants will be randomized to 3,330 mg/day Lysulin (1,110 mg tbl, TID) as add-on supplement therapy for 12 weeks. Follow-up visits will be at weeks 6 and week 12 (end of study). Baseline and follow-up visits will include physical examination, patient history and blood draw. The primary study outcome measure will be fasting plasma glucose and HbA1c. Secondary outcome measures will include fasting plasma C-peptide and AGE concentrations. A linear mixed effects model will be used to evaluate treatment-induced endpoints. The models will be fit for sequential values of the response variable (including the baseline measurement).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* HbA1c ≥7.5% and <10.0% within past 6 weeks on diet only or stable doses of oral antihyperglycemic agents with or without insulin
* stable body weight (< 5% change in last 3 months)
* If on insulin therapy: < 20% variation in insulin units 6 weeks prior to the study.

Exclusion Criteria:

* Type 1 DM
* current or recent use of supplements containing lysine, zinc or vitamin C
* uncontrolled hypertension (blood pressure ≥160/90 mmHg)
* kidney disease (serum creatinine GFR ≤50 mL/min)
* major illness
* severe gastrointestinal disease
* pregnancy
* liver function tests > 2.5 times normal values in the past 3 months
* currently abusing alcohol or drugs, or have a history of alcohol or drug abuse that in the investigator's opinion could cause the subject to be non-compliant; or have a general history of non-compliance with medications

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | Baseline
  Fasting plasma glucose
Fasting glucose | 6 weeks
  Fasting plasma glucose
Fasting glucose | 12 weeks
  Fasting plasma glucose
Hemoglobin A1c | Baseline
  Hemoglobin A1c measured by PVAHS pathology lab
Hemoglobin A1c | 12 weeks
  Hemoglobin A1c measured by PVAHS pathology lab

SECONDARY OUTCOMES:
Fasting C-peptide | Baseline
  Plasma C-peptide measured by ELISA
Fasting C-peptide | 12 weeks
  Plasma C-peptide measured by ELISA
CML | Baseline
  Nɛ-carboxymethyl lysine in plasma
CML | 12 weeks
  Nɛ-carboxymethyl lysine in plasma
CEL | Baseline
  Nɛ-carboxyethyl lysine in plasma
CEL | 12 weeks
  Nɛ-carboxyethyl lysine in plasma
GH1 | Baseline
  Glyoxal hydroimidazolone in plasma
GH1 | 12 weeks
  Glyoxal hydroimidazolone in plasma
3DGH1 | Baseline
  3-deoxyglucosone hydroimidazolone in plasma
3DGH1 | 12 weeks
  3-deoxyglucosone hydroimidazolone in plasma
MGH1 | Baseline
  Methylglyoxal hydroimidazolone in plasma
MGH1 | 12 weeks
  Methylglyoxal hydroimidazolone in plasma
MetSO | Baseline
  Methionine sulfoxide in plasma
MetSO | 12 weeks
  Methionine sulfoxide in plasma
2-AAA | Baseline
  2-aminoadipic acid in plasma
2-AAA | 12 weeks
  2-aminoadipic acid in plasma

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Phoenix VA Healthcare System, Phoenix, Arizona
  - Phoenix VA Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request. To protect the privacy and confidentiality of the research subjects, data will be de-identified by stripping all 18 HIPAA identifiers as comma-delimited text (.csv) files to ensure it is impossible to back out any changes and recover identifiable information.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3 years

DOCUMENTS (2):
  • Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT04234581/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT04234581/Prot_SAP_001.pdf